CLINICAL TRIAL: NCT06022679
Title: CBCT Analysis of the Craniofacial Architecture in Young, Non-overweight Apneic Adult Phenotype
Acronym: ACAS-3D
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Liege (Other)
Responsible Party: Principal Investigator, Jadoul Mathilde, post graduated dento facial orthopedic department, Centre Hospitalier Universitaire de Liege
Other Study IDs: B7072022000010; 2022/72 (Other: CHULiege)
Record Dates: First submitted 2023-08-16; First posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: OSA
Keywords: Young no-overweight adult; OSA; cephalometry; 3D

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test group SAHOS: The test group consisted of 23 patients ( 9 girls and 14 boys) recruited on the basis of polysomnography at sleep center of CHU Liege for suspected sleep disorders between 1 january 2022 and 1 april 2023, with IAH >15
  Interventions: Other: CBCT
- Control group no SAHOS: Concerning the control group, the participants, adults volunteers are recruited among friends and families of students who collaborate with sleep center for scientific projects. These subjects have no complaints related to OSA and will have to undergo a sleep examination (ventilatory polygraphy) to certify the absence of OSA. This group consisted of 23 patients (14 girls and 9 boys).
  Interventions: Other: CBCT

INTERVENTIONS:
Other: CBCT — CBCT examination in supine position A computerized 3D-analysis using Dolphin Imaging 11.95 software was performed in each CBCT.

SUMMARY:
This prospective, controlled study will compare the 3D cephalometric analysis of bone and craniofacial soft tissues in young (18-35 years) non-overweight apneic adults phenotype between a test group (with AHI 15) and a control group (healthy subjects with AHI < 15).

DETAILED DESCRIPTION:
Objectives The goal of this study is to determine an accurate bone and soft tissue phenotype for the non-overweight apneic young adult.

Materials and Methods This study was approved by the ethics medical committee of the University hospital of Liege.

This prospective, controlled study will compare cephalometric 3D analysis of bone and craniofacial soft tissue phenotype of young, non-overweight apneic adults using cephalometric 3D analysis between a test group (with AHI 15) and a control group (healthy subjects with AHI < 15).

The inclusion criteria were : (1) patients aged between 18 and 35 years ; (2) Body Mass Index (BMI) lower than 30kg/m² ; (3) alcohol consumption less than 4 unit per day ; (4) tabacco use less than 6 cigarettes per day ; (5) no illicit drug use ; and (6) absence of chronic pathology or medication.

The exclusion criteria were : (1) presence of an acute illness on the day of admission ; (2) patients treated with orthognathic surgery after apnea screening ; (3) patients with polysomnography with a sleep treatment device (PPCN or Mandibular advancement device).

The test group consisted of 23 patients (9 girls and 14 boys) recruited in polysomnography in sleep center of CHU Liege for suspected sleep disorders between 1 january 2022 and 1 april 2023.

Concerning the control group, the participants, healthy adults volunteers are recruited among friends and families of students who collaborate with sleep center for scientific projects. These subjects have no complaints related to OSA and will have to undergo a sleep examination (ventilatory polygraphy) to certify the absence of OSA. This group consisted of 23 patients (14 girls and 9 boys).

This study takes place in two stages. First, all patient are invited to an initial consultation where question about demographics (age, weight, height, gender) and medical history will be asked. At the end of this consultation, only patient of the control group leave with a sleep monitor to record their sleep for one night.

Afterwards, all patients (test and control group) will be invited to undergo a super low dose CBCT in the supine position at CHU Sart Tilman University Hospital.

Demographics and orthodontics data A general history will be taken, including gender, age, height, weight, medical and surgical history (e.g. presence/absence of tonsils and vegetations), current or past regular medication use, presence of allergies associated with allergic rhinitis, presence of asthma and presence of parafunctions.

Cephalometric data An ultra low dose CBCT ( 300μm resolution) will be performed in each patient with a field of 16x18 cm. A computerized 3D analysis will be performed with Dolphin Imaging 11.95 software. All these tools will allow the collection of the following data: parameters concerning the morphological typology and growth potential, the base of the skull, the maxilla, the mandible, the inter-maxillary relationship, the pharynx, the airways as well as the volumes of the different structures.

Sleep data The data will be collected by means of the epworth sleepiness scale (ESS) and a sleep recording of the polysomnography at the hospital type (AASM type 1 sleep recording) for the test group and of the ventilatory polygraph type (AASM type 3 sleep recording) for the control group.

ELIGIBILITY:
Inclusion Criteria:

* (1) patients aged between 18 and 35 years ;
* (2) Body Mass Index (BMI) lower than 30kg/m² ;
* (3) alcohol consumption less than 4 unit per day ;
* (4) tabacco use less than 6 cigarettes per day ;
* (5) no illicit drug use ; and
* (6) absence of chronic pathology or medication.

Exclusion Criteria:

* (1) presence of an acute illness on the day of admission ;
* (2) patients treated with orthognathic surgery after apnea screening ;
* (3) patients with polysomnography with a sleep treatment device (PPCN or Mandibular advancement device).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young people (18-35 years) non-overweight apneic divided into 2 groups: a test group (with AHI 15) and a control group (healthy subjects with AHI < 15).
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
maxillary volume | 2month
  maxillary volume with 3D cephalométric analysis

CONTACTS AND LOCATIONS:
Overall Officials: Annick AB Bruwier, Study Director — Service d'orthopédie dento-faciale CHU Liège; mathilde jadoul, Principal Investigator — Service Orthopédie dento-faciale CHU Liege
Locations (1):
- CHU Liège, site Brull, Liège, Belgium

REFERENCES:
- [Derived] Jadoul M, Albert A, Maes N, Poirrier R, Poirrier AL, Bruwier A. Three-dimensional cone beam computed tomography analysis of craniofacial phenotype in nonobese apneic young adults. Laryngoscope Investig Otolaryngol. 2025 Jan 31;10(1):e70061. doi: 10.1002/lio2.70061. eCollection 2025 Feb. PMID 39897118